CLINICAL TRIAL: NCT01254071
Title: An Open-label, Randomized, Single Dose, Two-Period Crossover Study to Determine the Bioavailability of a Fixed Dose Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.2mg) Relative to Co-administration of Dutasteride 0.5mg Capsules and Tamsulosin Hydrochloride 0.2mg
Brief Title: A Study to Determine the Bioavailability of a Fixed Dose Combination Product of Dutasteride (0.5mg) and Tamsulosin Hydrochloride (0.2mg) Relative to Co-administration of the Individual Components in Healthy Male Subjects of North East Asian and Non-Asian Ancestry.
Acronym: ARI114694
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 114694
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Prostatic Hyperplasia
Keywords: GI198745; Tamsulosin hydrochloride; Dutasteride; food effect; healthy male subjects; north-east Asian ancestry; Bioequivalence; cross-over design; Pilot bioequivalence
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fixed dose combination product (Experimental): Fixed Dose Combination capsule containing dutasteride 0.5mg and tamsulosin 0.2 mg
  Interventions: Drug: Dutasteride (0.5mg); Tamsulosin hydrochloride (0.2mg); fixed dose combination product of duatsteride (0.5mg) and tamsulosin hydrochloride (0.2mg)

INTERVENTIONS:
Drug: Dutasteride (0.5mg); Tamsulosin hydrochloride (0.2mg); fixed dose combination product of duatsteride (0.5mg) and tamsulosin hydrochloride (0.2mg) — In the first dosing session, twenty-two subjects of each cohort will receive the FDC capsule (dutasteride and tamsulosin hydrochloride (0.5mg/0.2mg) and the other 22 will receive commercial capsules of dutasteride 0.5mg and commercial tablets of tamsulosin hydrochloride 0.2mg co-administered. Following a wash-out period of at least 28 days, those subjects who received the FDC capsule in session 1, will be co-administered commercial capsules of dutasteride 0.5mg and commercial tablets of tamsulosin hydrochloride 0.2mg while those who were co-administered commercial capsules of dutasteride 0.5mg and commercial tablets of tamsulosin hydrochloride 0.2mg in session 1 will receive the FDC capsule in the second dosing session.

SUMMARY:
This study will be an open-label, randomized, single dose, two-period crossover study to determine the bioavailability of a fixed dose combination capsule formulation of dutasteride and tamsulosin hydrochloride (0.5mg/0.2mg) relative to co-administration of dutasteride 0.5mg capsules and tamsulosin hydrochloride 0.2mg tablets in healthy male subjects of North East Asian and non-Asian ancestry. Subjects will receive single oral doses of a combination capsule formulation of dutasteride 0.5 mg/ tamsulosin 0.2 mg in a fed or fasted state or concomitant dosing of dutasteride 0.5 mg and the Japan-sourced Harnal-D 0.2 mg in a fed or fasted state. Each dose of study medication will be separated by a 28-day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate, safety laboratory data, and review of adverse events. The study will enrol 88 healthy male subjects to ensure that 80 complete the study. At least twenty percent of the study population will be of Japanese ancestry, approximately 20% will be of Chinese ancestry and approximately 20% of Korean ancestry while the remainder of the population will be of non-Asian ancestry.

DETAILED DESCRIPTION:
Description:

This study will be an open-label, randomized, single dose, two-period crossover study to determine the bioavailability of a fixed dose combination capsule formulation of dutasteride and tamsulosin hydrochloride (0.5mg/0.2mg) relative to co-administration of dutasteride 0.5mg capsules and tamsulosin hydrochloride 0.2mg tablets in healthy male subjects of North East Asian and non-Asian ancestry. Subjects will receive single oral doses of a combination capsule formulation of dutasteride 0.5 mg/ tamsulosin 0.2 mg in a fed or fasted state or concomitant dosing of dutasteride 0.5 mg and the Japan-sourced Harnal-D 0.2 mg in a fed or fasted state. Each dose of study medication will be separated by a 28-day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate, safety laboratory data, and review of adverse events. The study will enrol 88 healthy male subjects to ensure that 80 complete the study. At least twenty percent of the study population will be of Japanese ancestry, approximately 20% will be of Chinese ancestry and approximately 20% of Korean ancestry while the remainder of the population will be of non-Asian ancestry.

Background:

Dutasteride (AVODART ™) is an approved potent 5-alpha-reductase inhibitor indicated for the treatment of symptomatic benign prostatic hyperplasia (BPH) in men with an enlarged prostate to improve symptoms, reduce the risk of acute urinary retention and reduce the risk of the need for BPH-related surgery [AVODART Package Insert, 2009].

In humans, dutasteride is well-tolerated in single doses up to 40mg/day, multiple doses up to 40mg/day administered for 7 days, and 5mg/day administered for 24 weeks. In clinical studies, the overall incidence and type of adverse events (AEs) was similar across the dutasteride, placebo, and finasteride treatment groups.

Tamsulosin (Harnal, Harnal D, Flomax) is an alpha-1-adrenoceptor blocking agent approved for the treatment of signs and symptoms of benign prostatic hyperplasia. Tamsulosin HCl is extensively metabolized, with less than 10% of the dose excreted in the urine unchanged [Harnal, 2009a; Harnal, 2009b; Flomax, 2009]. In human liver microsomes and human lymphoblastoid cells expressing CYP cDNAs in vitro, tamsulosin HCl is metabolized by both CYP3A4 and CYP2D6 [Matsushima, 1998].

Clinical data exist to support that tamsulosin (an alpha-1-adrenoceptor antagonist), when used in combination with dutasteride (a 5-alpha reductase inhibitor), offers a more effective treatment for the symptoms of benign prostatic hyperplasia than either drug used alone [GSK study ARI40005, GlaxoSmithKline document number HM2002/00171/01]. In addition, data from a large, multi-centre National Institutes of Health-sponsored Medical Therapy of Prostatic Symptoms (MTOPS) study revealed greater benefits of combination alpha-1-adreoceptor antagonist and 5-alpha-reductase inhibitor therapy compared with either monotherapy in males with BPH [McConnell, 2002].

Clinical drug interaction studies have shown no pharmacokinetic or pharmacodynamic interactions between dutasteride and tamsulosin. Dutasteride may be administered with or without food. Tamsulosin should be administered with food. While there is food effect PK data on dutasteride and tamsulosin when administered individually, an objective of this study is to evaluate the effect of food (high fat meal state versus fasted state) on the absorption of dutasteride and tamsulosin HCl when given in a combination capsule formulation relative to the co-administration of the two components, dutasteride and tamsulosin HCl. A previous study, ARI109882, [GlaxoSmithKline document number ZM2007/00022/00], also determined the bioequivalence and food effect of the combination capsule formulation relative to the co-administration of each component administered separately. In that study, the GSK combination capsule was found to be bioequivalent (under both fed and fasted conditions) to the marketed products administered separately. In the present study, the dose of tamsulosin HCl administered will be lower than in ARI109882 (0.2 mg versus 0.4mg administered in ARI109882). The dose of dutasteride is the same in both studies (0.5mg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Males between 20 and 45 years of age inclusive, at the time of signing the informed consent form.
* Japanese ancestry defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese, or Korean ancestry defined as being born in Korea, having four ethnic Korean grandparents, holding a Korean passport or identity papers and being able to speak Korean, or Chinese ancestry defined as being born in China, Hong Kong, Singapore or Taiwan, having four ethnic Chinese grandparents, holding a Chinese passport or identity papers and being able to speak Chinese.

Japanese, Korean and Chinese subjects should also have lived outside their respective countries for less than 10 years.

* Male subjects with female partners who are either pregnant or suspected of being pregnant must agree to the use of a condom during sexual activity. This criterion must be followed from the time of the first dose of study medication until 28 days after the last dose of study medication.
* BMI : For Caucasians: BMI within the range 18 -30 kg/m2 (inclusive); weight range 55-95 kg (inclusive) For East Asians: BMI within the range 18 -28 kg/m2 (inclusive) and height 1.55m-1.85m (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcB < 450 msec.
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

Medical Conditions Exclusions:

* Poor metabolizer for CYP2D6 substrates as determined by genotyping of selected CYP2D6 variants at screening.
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* Subject is mentally or legally incapacitated.

Medication Exclusions:

* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort, Black Khosh, Dong Quai, Milk Thistle, licorice) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to tamsulosin hydrochloride or durasteride, components thereof or drugs of this class or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Lifestyle Exclusions:

* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the screening visit defined by the following Australian guidelines:

Males: An average weekly intake greater than 21 units or an average daily intake greater than 3 units. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits and 100 mL of wine.

Subjects must be able and willing to abstain from beverages and foods containing alcohol 24 hours prior to and during the dosing day.

* Consumption of red wine, grapefruit juice, grapefruit and related hybrids, jufen grapes from 7 days prior to the first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2010-09-10 (Actual); Primary Completion 2010-12-21 (Actual); Study Completion 2010-12-21 (Actual)

PRIMARY OUTCOMES:
1. To investigate the bioavailability of a combination capsule formulation of dutasteride 0.5 mg/ tamsulosin HCl 0.2 mg relative to concomitant dosing of dutasteride 0.5 mg capsules and tamsulosin 0.2 mg tablets in the fed and fasted states. | PK at pre-dose, at 15,30 and 45 min; 1, 2,3,4,6,8,10,12,16,24,48,and 72 hours.

SECONDARY OUTCOMES:
1. To investigate the effect of food on the bioavailability of a combination capsule formulation of dutasteride 0.5 mg/ tamsulosin HCl 0.2 mg relative to concomitant dosing of dutasteride 0.5 mg capsules and tamsulosin 0.2 mg tablets. | PK at pre-dose, 15, 30,and 45 mins; 1,2,3,4,6,8,10,12,16,24,48,and 72 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Flomax (Tamsulosin hydrochloride) Product Information for the USA, 2009
- [Background] GlaxoSmithKline Document Number ZM2007/00022/00. ARI109882. An Open-Label, Randomized, Single Dose, Three-Period Crossover Study to Determine the Bioequivalence and Food Effect of a Combination Capsule Formulation of Dutasteride and Tamsulosin Hydrochloride (0.5mg/0.4mg) Compared to Concomitant Dosing of AVODART 0.5mg and Flomax 0.4mg Commercial Capsules in Healthy Male Subjects, August 2007
- [Background] GlaxoSmithKline studyARI40005: A randomised, double-blind, parallel group study to investigate the efficacy and safety of treatment with Dutasteride (0.5mg) and Tamsulosin (0.4mg), administered once daily for 4 years, alone and in combination, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic benign prostatic hyperplasia; [GlaxoSmithKline Document Number HM2002/00171/01].
- [Background] Harnal capsule (Tamsulosin hydrochloride), 0.4mg Product Information for Australia, 2009b.
- [Background] Harnal D (Tamsulosin hydrochloride), extended release tablet, 0.2mg Product Information for Hong Kong, 2009a.
- [Background] Matsushima H, Kamimura H, Soeishi Y, Watanabe T, Higuchi S, Tsunoo M. Pharmacokinetics and plasma protein binding of tamsulosin hydrochloride in rats, dogs, and humans. Drug Metab Dispos. 1998 Mar;26(3):240-5. PMID 9492387
- [Background] McConnell JD. The long term effects of medical therapy on the progression of BPH: Results from the MTOPS Trial (abstract 1042). J. Urology 167 (4):265, 2002.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114694 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114694?search=study&search_terms=114694#rs
- Available data/document: Study Protocol: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114694 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register